CLINICAL TRIAL: NCT00408447
Title: Allogeneic Stem Cell Transplant to Induce Mixed Donor Chimerism in Patients With Sickle Cell Disease and Thalassemia
Brief Title: Stem Cell Transplant in Sickle Cell Disease and Thalassemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Monica Bhatia, Professor of Pediatrics, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA7701; CHNY-01-503 (Other: CU)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Beta Thalassemia
Keywords: stem cell transplant; sickle cell disease; thalassemia; moderately ablative; cord blood transplant; matched family donor
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; Thalassemia | interventions — Busulfan; fludarabine; fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCD group (Other): Sickle Cell Disease patients receiving chemotherapy (Busulfan, Fludarabine and Alemtuzumab) will undergo allogeneic stem cell transplant.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Alemtuzumab; Procedure: Allogeneic stem cell transplant
- BT group (Other): Beta Thalassemia patients receiving chemotherapy (Busulfan, Fludarabine and Alemtuzumab) will undergo allogeneic stem cell transplant.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Alemtuzumab; Procedure: Allogeneic stem cell transplant

INTERVENTIONS:
Drug: Busulfan — Busulfan 4 mg/kg/d x 4d
  Other Names: Busulfex
Drug: Fludarabine — Fludarabine 30 mg/m2/d x 6d
  Other Names: Fludara
Drug: Alemtuzumab — Alemtuzumab 2mg/m2 x 1d, 6mg/m2 x 2 d, 20mg/m2 x 2d
  Other Names: Campath
Procedure: Allogeneic stem cell transplant — Allogeneic stem cells will be given on day 0 (after chemotherapy conditioning)obtained either from a family donor (first degree relative) or sibling cord blood donor.
  Other Names: Related Bone Marrow; Related Cord Blood

SUMMARY:
The primary purpose of this study is to see if giving lower doses of chemotherapy (moderately ablative) will result in successful bone marrow replacement without as severe side-effects but with permanent control of the disease. Patients will receive a chemotherapy regimen with busulfan, fludarabine, and alemtuzumab followed by an infusion of stem cells, either from a family-related or cord-blood matched donor.

DETAILED DESCRIPTION:
Sickle cell disease is a genetic disorder in which a mutation in the beta chain of human hemoglobin results in abnormal blood hemoglobin, causing red blood cells to sickle under stress with resulting symptoms including severe pains and strokes. Beta thalassemia is another genetic disorder in which there are abnormal beta hemoglobin chains, causing anemia. In both disorders, frequent red blood cell transfusions may be required to sustain life, but these often result in complications including multiple hospitalizations, iron overload, or bacterial or viral infections such as hepatitis. Standard drugs and therapies used in the treatment of sickle cell disease and/or beta thalassemia provide only supportive care, and may result in long-term side effects, and inadequate control of the disease process. Bone marrow transplant has been increasingly used for the long-term treatment and cure of sickle cell disease and beta thalassemia. Although, not without acute and potential long term side effects, this alternative offers long term control and potential cure of the disease. Most of the side effects seen with bone marrow transplant are directly related to the high intensity of chemotherapy used (ablative).

ELIGIBILITY:
Inclusion Criteria:

Sickle Cell Disease:

* Diagnosis of Homozygous Hemoglobin S Disease or Heterozygous Hemoglobin Sickle Cell (SC) or S 0/+ thalassemia, or Sickle/variant resulting in Chronic Hemolytic Anemia with hemoglobin (HgB) ≤10 mg/dL
* Age ≤30
* Matched sibling donor and asymptomatic, or 8/8 human leukocyte antigen (HLA) matched unrelated adult donor

Patient must have adequate organ function as below:

* Adequate renal function defined as serum creatinine ≤1.5 x normal, or Creatinine clearance or radioisotope glomerular filtration rate (GFR) >100 ml/min/1.73 m2 or >70ml/min/1.73m2 for patients >16 years old
* Adequate liver function defined as serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase (ALT)) < 5.0 x normal
* Adequate Cardiac Function defined as shortening fraction of ≥28% by echocardiogram, or ejection fraction of ≥48% by radionuclide angiogram or echocardiogram
* Adequate pulmonary function defined as corrected Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% by pulmonary function test, or for children who are unable to perform DLCO maneuver ≥85% O2 saturation, no evidence of dyspnea at rest

Exclusion criteria:

General

* Karnofsky/Lansky Performance Score <60%
* Demonstrated lack of compliance with medical care
* Pregnant or nursing
* Evidence of uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms) within 1 month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.

Histologic Exam of Liver (liver biopsy) with bridging fibrosis or cirrhosis.

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of toxicity associated with moderately ablative therapy (busulfan/fludarabine/alemtuzumab) and allogeneic stem cell transplantation in selected patients with Sickle Cell Disease (SCD) and Beta Thalassemia (BT) | Day 30, Day 60, Day 100, Day 180, 1 year, 2 years, 3 years, 5 years, 10 years
  To examine if giving lower doses of chemotherapy will result in less severe side-effects but with permanent control of the disease.

SECONDARY OUTCOMES:
Time to donor hematological reconstitution (neutrophil, red blood cell and platelet recovery) following moderately ablative therapy and allogeneic stem cell transplantation in selected patients with SCD and BT | days 60, 100, 180, 365, 730
  To examine if giving lower doses of chemotherapy and bone marrow replacement can result in control of the disease.
Incidence of acute and chronic graft versus host disease (GVHD) following moderately ablative therapy and allogeneic stem cell transplantation in selected patients with SCD and BT | as clinically appropriate
  To examine if giving lower doses of chemotherapy will result in successful bone marrow replacement.
Percent of patients who have either a complete, very good partial, partial or no response (clinical/laboratory) following moderately ablative therapy and allogeneic stem cell transplantation in selected patients with SCD and BT | 6mos, 1 yr, 2 yr
  To examine if giving lower doses of chemotherapy with bone marrow replacement will result in good control of the disease.
Quality of life (QOL) score | Day +180; year 1, 3, 5, 10
  To determine the impact of moderately ablative stem cell transplant on quality of life and neurocognitive functioning with SCD over time
Incidence of primary and secondary graft failure | Day +42, +60,
  To collect data on graft failure
Percent of mixed donor chimerism | Day +30, 60, 100, 180, 365, 730, and 1005
  To collect data on donor chimerism

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bhatia, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York-Presbyterian, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Satwani P, Harrison L, Morris E, Del Toro G, Cairo MS. Reduced-intensity allogeneic stem cell transplantation in adults and children with malignant and nonmalignant diseases: end of the beginning and future challenges. Biol Blood Marrow Transplant. 2005 Jun;11(6):403-22. doi: 10.1016/j.bbmt.2005.04.002. PMID 15931629
- [Background] Del Toro G, Satwani P, Harrison L, Cheung YK, Brigid Bradley M, George D, Yamashiro DJ, Garvin J, Skerrett D, Bessmertny O, Wolownik K, Wischhover C, van de Ven C, Cairo MS. A pilot study of reduced intensity conditioning and allogeneic stem cell transplantation from unrelated cord blood and matched family donors in children and adolescent recipients. Bone Marrow Transplant. 2004 Mar;33(6):613-22. doi: 10.1038/sj.bmt.1704399. PMID 14730337
- [Derived] Bhatia M, Jin Z, Baker C, Geyer MB, Radhakrishnan K, Morris E, Satwani P, George D, Garvin J, Del Toro G, Zuckerman W, Lee MT, Licursi M, Hawks R, Smilow E, Baxter-Lowe LA, Schwartz J, Cairo MS. Reduced toxicity, myeloablative conditioning with BU, fludarabine, alemtuzumab and SCT from sibling donors in children with sickle cell disease. Bone Marrow Transplant. 2014 Jul;49(7):913-20. doi: 10.1038/bmt.2014.84. Epub 2014 May 5. PMID 24797180